CLINICAL TRIAL: NCT04519372
Title: SARS-CoV-2 /COVID-19 Admission Screening in a University Hospital Setting (Covid-Screen Quality Control Study)
Brief Title: SARS-CoV-2 /COVID-19 Admission Screening in a University Hospital Setting
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-00808
Record Dates: First submitted 2020-08-17; First posted 2020-08-19 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Covid19; SARS-CoV-2
Keywords: Screening; asymptomatic
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Testing for SARS-CoV-2 — All Patients admitted to the hospital were routinely tested for SARS-CoV-2 within 72 hours of admission by nasopharyngeal swabs.

SUMMARY:
The proportion of asymptomatic carriers of SARS-CoV-2 remains elusive, so the potential benefit of systematic screening during the SARS-CoV-2-pandemic is controversial. We investigate the proportion of asymptomatic inpatients who were identified by systematic screening for SARS-CoV-2 upon hospital admission.

Adult patients admitted to the University Hospital Basel from 01.04.-14.06.2020 were routinely tested for SARS-CoV-2 within 72 hours of admission by nasopharyngeal swabs.

Each patient screened during the study period was retrospectively classified symptomatic or asymptomatic for COVID-19 based on medical chart review.

ELIGIBILITY:
Inclusion Criteria:

* The patient population is defined as all adult patients hospitalized in the University Hospital Basel from April 1st, 2020 to June 14th, 2020.

Exclusion Criteria:

* Outpatients
* Patients with SARS-CoV-2 screening in the outpatient test center
* Patients with a SARS-CoV-2 test more than 72 hours before hospital admission
* Test not performed (for any reason)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population is defined as all patients with an inhospital casenumber and a screening swab for SARS-CoV-2 at the University Hospital Basel from April 1st, 2020 to June 14th, 2020.
Sampling Method: Non-Probability Sample
Enrollment: 4099 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-06-14 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Proportion of SARS-CoV-2 -infected patients | 01.04.2020-14.06.2020
  We aim to determine the proportion of SARS-CoV-2-infected patients detected by systematic at-admission screening

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Tschudin-Sutter, Prof. Dr. MD, Principal Investigator — University Hospital Basel, Division of Infectious Diseases and Hospital Epidemiology
Locations (1):
- University Hospital Basel, Division of Infectious Diseases and Hospital Epidemiology, Basel, Switzerland